CLINICAL TRIAL: NCT02235129
Title: Six Minute Walking Test and Breath-holding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 6MWTBH
Record Dates: First submitted 2014-07-24; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breath Holding

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- 6 minutes walking test (Experimental)
  Interventions: Other: breath-holding

INTERVENTIONS:
Other: breath-holding

SUMMARY:
To compare the relationship between breath-hold time and the distance in a Six Minute Walking Test in chronic obstructive pulmonary disease population.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic obstructive pulmonary disease

Exclusion Criteria:

* contra-indication for six minutes walking test
* difficulty to walk
* musculoskeletal disorder

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
six minute walking test | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium